CLINICAL TRIAL: NCT04386759
Title: COVID-19 Infection in Healthcare Workers: a Cohort Study
Brief Title: COVID-19 Infection in Healthcare Workers
Acronym: HOP-COVID
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200483
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: COVID-19; Healthcare workers; Incidence; Risk factors; Nosocomial infection
MeSH Terms: conditions — COVID-19; Cross Infection | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Up to protocol v2.0: Filling when including a first self-survey concerning the period of the last fifteen days. The following questionnaires will be completed online every week until the end of the study. For healthcare worker who have already presented a symptomatic infection at the time of inclusion, only the self-survey "inclusion" will be completed, it will relate to the period of fifteen days preceding the diagnosis.
  From protocol v3.0: After performing a RT-PCR or an antigenic test for COVID diagnosis, the healthcare workers will complete a unique self-questionnaire about individual and contextual risks factors during the 15 days preceding the test.
  Interventions: Other: Cohort

INTERVENTIONS:
Other: Cohort — None. Only implementation of a cohort with data collection via individual self-questionnaires and administrative services for contextual data.

SUMMARY:
Introduction: The SARS-Cov-2 outbreak in France and the concomitant massive increase in the number of cases requiring hospital management create a major risk of COVID-19 infection for hospital staff. In addition to nosocomial transmission, the health care workers (HCWs), defined as persons serving in health care settings who have the potential for direct or indirect exposure to patients or infectious materials, are also exposed to community transmission. Whether HCWs acquire infection at work or in the community is important to adapt protection measures. A few studies investigated COVID-19 infection among medical and nursing personnel. However, none have analyzed all categories of hospital staff. As of April 9, 2020, a total of 9,282 US HCWs with confirmed COVID-19 had been reported to CDC (US), however description of occupational activities was not available. Therefore, limited information is available about COVID-19 infection among HCWs.

Thus, the objectives of the sdudy are to estimate the incidence of symptomatic SARS-CoV-2 infection in HCWs in five university hospitals (including geriatric hospitals) of the great Paris area and to estimate both nosocomial and community risk factors.

Method: A prospective and retrospective cohort study that includes all hospital staff (including medical and nursing personnel, health care managers, laboratory, radiology, reception staffs, stretcher-bearers, etc.) working in different departments of five university hospitals (acute medical centers and geriatric hospitals) in the great Paris area (9 000 HCWs). Incidence of symptomatic SARS-CoV-2 infection will be estimated with its 95%CI. Individual and contextual risk factors will be analyzed using multilevel multivariate logistic regression modelling to account for clustering and confounding.

Conclusion This study should make it possible to better characterize SARS-Cov-2 contamination of HCWs and to estimate the share of nosocomial transmission.

DETAILED DESCRIPTION:
Details for "Study design" section

Time perspective : Retrospective and prospective cohort study.

Up to protocol v2.0: Data from healthcare workers with COVID+ diagnostic at the time of inclusion will only be collected retrospectively. In contrast, data from healthcare workers free from infection will be collected prospectively.

From protocol v3.0: Recruitment of healthcare workers will be prospective. A retrospective collection of exposures during the 15 days preceding the RT-PCR or the antigenic test for COVID diagnosis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff working in any of the 5 hospitals participating in the study,
* Of legal age,
* With or without a previous diagnosis of COVID-19 infection,
* Patient with a SARS-CoV-2 screening by RT-PCR or antigenic test (from version 3.0 of the protocol)
* Not opposed to participating in the research

Exclusion Criteria:

* Unable or unwilling to complete the non-opposition
* Unable or unwilling to complete an online self-questionnaire (eCRF)
* Opposition to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults healthcare workers, who are not opposed to participating in research.
Sampling Method: Non-Probability Sample
Enrollment: 1858 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
SARS-COV-2 infection | Up to 3 months
  The primary endpoint will be the occurrence of confirmed (RT-PCR or antigenic test or work stopping) SARS-CoV-2 infection.

SECONDARY OUTCOMES:
SARS-COV-2 incidence regarding hospitals, assigned services and profession | Up to 3 months maximum
  Information collected by a self questionnaire and service datas
Individual and contextual risks factors | Up to 3 months maximum
  Risks factor are collected by a self questionnaire and service datas

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BASTUJI-GARIN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
Datas are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information.

REFERENCES:
- [Derived] Bastuji-Garin S, Brouard L, Bourgeon-Ghittori I, Zebachi S, Boutin E, Hemery F, Fourreau F, Oubaya N, De Roux Q, Mongardon N, Fourati S, Decousser JW. The Relative Contributions of Occupational and Community Risk Factors for COVID-19 among Hospital Workers: The HOP-COVID Cohort Study. J Clin Med. 2023 Feb 2;12(3):1208. doi: 10.3390/jcm12031208. PMID 36769854